CLINICAL TRIAL: NCT03774628
Title: Long-term Immunity of Rabies Vaccine(Human Diploid Cell)for Human Use,Freeze-dried and Booster Dose Effects at 10 Years Post-primary Vaccination
Brief Title: Immunity Duration of Rabies Vaccine and Booster Dose Effects at 10 Years Post-primary Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT061
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chengdu Kanghua (one booster shot) (Experimental): one dose, A rabies vaccine (human diploid cell) for human use, Freeze-dried produced by Chengdu Kanghua Biological Products Co.,Ltd.
  Interventions: Biological: Chengdu Kanghua (one booster shot)
- Chengdu Kanghua (two booster shots) (Experimental): two doses at 0 and 3 days, on A rabies vaccine (human diploid cell) for human use, Freeze-dried produced by Chengdu Kanghua Biological Products Co.,Ltd.
  Interventions: Biological: Chengdu Kanghua (two booster shots)

INTERVENTIONS:
Biological: Chengdu Kanghua (one booster shot) — A rabies vaccine (human diploid cell) for human use, Freeze-dried produced by Chengdu Kanghua Biological Products Co.,Ltd. 1.0 ml experimental vaccine on day 0
  Arms: Chengdu Kanghua (one booster shot)
Biological: Chengdu Kanghua (two booster shots) — A rabies vaccine (human diploid cell) for human use, Freeze-dried produced by Chengdu Kanghua Biological Products Co.,Ltd. 1.0 ml experimental vaccine on day 0 and 3
  Arms: Chengdu Kanghua (two booster shots)

SUMMARY:
A rabies vaccine (human diploid cell) for human use, Freeze-dried produced by Chengdu Kanghua Biological Products Co.,Ltd is used to prevent human rabies. The vaccine was completed in the Phase III clinical trial from August 2008 to February 2009 in Lianshui County, Jiangsu Province (Approval of Drug Clinical Trial No. 2008L03156). A total of 1200 subjects aged 10-60 years were randomly assigned trial group (Kanghua vaccine group, 600 participants) and control groups (Pasteur vaccine group, 600 participants). The result showed that this vaccine could provide good immunogenicity and mild adverse reactions. On April 28, 2012, the drug registration approval was obtained (Approval No. 2012S00222).

To disclose the effects of booster immunization of human diploid cell rabies vaccine (HDCV) after eight years of primary vaccination. Sixty subjects who had participated the phase Ⅲ clinical trial of freeze-dried HDCV were selected and given booster immunization after eight years of primary vaccination. The result showed that the freeze-dried HDCV has good immune effects with one-dose of booster immunization after eight years of primary vaccination． In order to find a ten years of immunization persistence and booster dose immune effect, the investigators decided to perform this immunization persistence and booster immunity trial among these subjects who had received five doses of rabies vaccine vaccines (around ten years after the fundamental immunity). The investigators do the recruitment among these subjects who had participated in the previous phase Ⅲ trail and the subjects were divided into two layers, such as trial group (Kanghua vaccine group) and the control group (Paste vaccine group). Each layer of the subjects randomly received one booster dose (Day 0) and two booster doses (Day 0, 3) the freeze-dried HDCV in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in the Phase III clinical study of the vaccine and completed the full immunization
* Subjects or legal guardians can and will comply with the requirements of the protocol
* Subjects are able to understand and sign the informed consent
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Female in pregnancy
* Subjects who have been vaccinated other rabies vaccines after participating in the phase III clinical study of the vaccine (excluding those who participated in the 8-year booster immunization)
* Subject who has serious adverse reaction history after vaccination such as allergies, hives, difficulty in breathing, angioedema or abdominal pain or allergic to any ingredient of the this rabies vaccine, including excipient
* Any acute disease, serious chronic disease, fever，and chronic disease at acute stage
* Subject with autoimmune diseases or immunodeficiency
* Subject with asthma, unstable over the past two years requiring emergency treatment, hospitalization, intubation, oral or intravenous corticosteroids
* Subject with diabetes (Type I or II) excluding gestational diabetes
* Subject with thyroidectomy history, or require treatment in the past 12 months due to thyroid disease
* Subject with coagulation abnormalities diagnosed by doctors (such as clotting factor deficiency, coagulation disorders, platelet disorder) or obvious bruises or blood clotting disorder
* Subject with cancer, or has been treated in active cancer period or not clearly cured, or may recur during the study period
* Subject with uncontrolled epilepsy or other progressive neurological disease
* Asplenia, functional asplenia, without a spleen or removal of the spleen caused by any situation
* Any prior administration of immunodepressant, cytotoxic treatment or inhaled corticosteroids in last 6 months, excluding those corticosteroid spray therapy for allergic rhinitis, topical corticosteroid treatment for acute non-concurrent dermatitis)
* Ongoing anti-tuberculosis prevention or treatment
* Subject who cannot comply with the trial requirements, or with mental illness/dual-stage affective psychosis in the past or at present
* Any medical, psychological, social or other condition judged by investigator, that may interfere subject's compliance with the protocol or signature on informed consent
* Untolerable adverse reactions occurred after booster dose injection within 10 years later;
* Any condition that in the opinion of the investigators may be not suitable for continued participation after booster dose injection within 10 years later

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Proportion of serum rabies virus neutralizing antibodies to protective levels 10 years after primary vaccination | 10 years after primary vaccination
  calculate the proportion of serum rabies virus neutralizing antibodies to protective levels 10 years after primary vaccination
Geometric mean concentration (GMC) of serum rabies virus neutralizing antibody 10 years after primary vaccination | 10 years after primary vaccination
  calculate the geometric mean concentration (GMC) of serum rabies virus neutralizing antibody 10 years after primary vaccination
Proportion of serum rabies virus neutralizing antibodies to protective levels | 6 hours, 1 day, 3 days, 7 days or 14 days after booster dose injection within 10 years later
  calculate the proportion of serum rabies virus neutralizing antibodies to protective levels 6 hours, 1 day, 3 days, 7 days or 14 days after booster dose injection within 10 years later
Positive seroconversion rate of serum rabies virus neutralizing antibody | 6 hours, 1 day, 3 days, 7 days or 14 days after booster dose injection within 10 years later
  calculate the positive seroconversion rate of serum rabies virus neutralizing antibody 6 hours, 1 day, 3 days, 7 days or 14 days after booster dose injection within 10 years later
Geometric mean concentration (GMC) of serum rabies virus neutralizing antibody | 6 hours, 1 day, 3 days, 7 days or 14 days after booster dose injection within 10 years later
  calculate the geometric mean concentration (GMC) of serum rabies virus neutralizing antibody 6 hours, 1 day, 3 days, 7 days or 14 days after booster dose injection within 10 years later
Mean geometric increases (GMIs) of serum rabies virus neutralizing antibody | 6 hours, 1 day, 3 days, 7 days or 14 days after booster dose injection within 10 years later
  calculate the mean geometric increases (GMIs) of serum rabies virus neutralizing antibody 6 hours, 1 day, 3 days, 7 days or 14 days after booster dose injection within 10 years later

CONTACTS AND LOCATIONS:
Locations (1):
- Lianshui Xinyi Center for Disease Control and Prevention, Huai'an, Jiangsu, China

REFERENCES:
- [Derived] Hu J, Wang S, Zhou R, Liu H, Gan X, Wei M, Zhu F, Meng F, Hou W. Long-term immunity and the effect of one or two booster doses with a lyophilized human rabies vaccine (human diploid cells) at 10 years post primary vaccination in China. Hum Vaccin Immunother. 2021 Sep 2;17(9):3162-3168. doi: 10.1080/21645515.2021.1906601. Epub 2021 May 4. PMID 33945439